CLINICAL TRIAL: NCT03178656
Title: RCT Research: the Treatment of Hepatic Carcinoma With Portal Vein Branch Tumor Thrombosis (Resection or Sorafenib)
Brief Title: A Trial to Compare Surgery With Sorafenib for Hepatic Celluler Cancer With Portal Vein Tumor Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: chenxp007
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Portal Vein Tumor Thrombus
Keywords: sorafenib, operation
MeSH Terms: interventions — Sorafenib; Surgical Procedures, Operative; TNF-Related Apoptosis-Inducing Ligand

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVTT WITH SORAFENIB (Active Comparator): AASLD recommend therapy:
  sorafenib tablet, 400mg, bid.
  Interventions: Drug: Sorafenib
- PVTT WITH OPERATION (Experimental): patients suitable for surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Drug: Sorafenib — continuous application of the drugs
  Other Names: control
  Arms: PVTT WITH SORAFENIB
Procedure: surgery — curative resection
  Other Names: trail
  Arms: PVTT WITH OPERATION

SUMMARY:
According to the guidelines recommended, only a few new targeted therapy drugs treatment, such as Sorafenib, is proper. It's 3 year survival rate is only 8% or so. According to our previous study, patients with hepatic carcinoma without portal vein tumor thrombus backbone and the contralateral tumor thrombus applyed tumor excision, along with tumor thrombus, the 3 year survival rate can reach 39.9%, the 5-year survival rate can reach 22.7%, curative effect is obviously better.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of Hepatic cellular Carcinoma. 2. Patients with Portal Vein Tumor Thrombus (PVTT) of Hepatic cellular Carcinoma (HCC) detected by Serum Alpha Fetoprotein (AFP) and CT or MRI.

  3. Patients with a solitary tumor or multiple tumor which are resectable. 4. Patients without Hepatic vein or bile duct invasion and extrahepatic metastasis.

  5. Patients without surgical contraindication. 6. Patients with Child A or B liver function and indocyanine green retention rate at 15min (ICGR15) < 10% before treatment.

  7. Laboratory examination: haemoglobin (Hb)>100g/L, white blood cell (WBC) > 3000/mL, PLT > 8×10*10/L before treatment.

  8. Patients without severe esophagealgastric varices before treatment. 9. Patients with HBV，HBV DNA≤100, 000 copy/mL. 10. All of the patients has written consent for this research.

Exclusion Criteria:

* 1.Patients with multiple tumors or vascular or bile duct invasion or extrahepatic metastasis.

  2.Patients with surgical contraindication. 3.Patients with Child C grade liver function before treatment. 4.Patients with other malignancy. 5.Patients treated with hepatic resection or TACE before this treatment. 6.Patients with severe esophagealgastric varices or refractory ascites or coagulation dysfunction before treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-04-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
overall survival of 1 year | 1 years
  including 3, 6, and 12 months overall survival (OS) rate
overall survival of 3 year | 3 years
  including 1, 2, and 3 years overall survival (OS) rate

SECONDARY OUTCOMES:
time to progression | 3 years
  deterioration indicated by complications or metastasis detected by CT, MRI and laboratory examination.

OTHER OUTCOMES:
mortality | 30 days
  death within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatic surgery center, Tong ji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No